CLINICAL TRIAL: NCT01390727
Title: Effects of Slow Breathing on Blood Pressure and Autonomic Function in Hypertensive Patients
Brief Title: Effects of Slow Breathing on Blood Pressure and Autonomic Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Decio Mion Jr., MD, Phd, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAPESP 2010/06921-2
Record Dates: First submitted 2011-05-23; First posted 2011-07-11 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Hypertension
Keywords: hypertension; device-guided breathing; autonomic function; Resperate
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Listen music (Placebo Comparator): After randomization, the patients allocated in this arm will be instructed to listen to calm music for 15 minutes per day during 8 weeks
  Interventions: Other: Listen music
- Device-guided breathing (Active Comparator): After randomization, the patients allocated in this arm will be instructed to use a device-guided breathing, for 15 minutes per day during 8 weeks, with the aim to reduce the respiratory frequency to less than 10 breaths/min
  Interventions: Device: Device-guided breathing (Resperate - InterCure, Israel)

INTERVENTIONS:
Device: Device-guided breathing (Resperate - InterCure, Israel) — After randomization, the patients allocated in this arm will be instructed to use a device-guided breathing, for 15 minutes per day during 8 weeks, with the aim to reduce the respiratory frequency to less than 10 breaths/min
  Arms: Device-guided breathing
Other: Listen music — After randomization, the patients allocated in this arm will be instructed to listen to calm music for 15 minutes per day during 8 weeks
  Arms: Listen music

SUMMARY:
Hypertension is a chronic disease that affects about 23% of the brazilian population. The treatment of hypertension by pharmacological intervention is efficacious, but has side effects and significant costs. Techniques that reduce the respiratory rate are shown as a effective non-pharmacological treatment in controlling blood pressure. Evidence has shown that a slow and deep breathing rate, around 10 breaths per minute or less, significantly reduces blood pressure. However, the physiological mechanisms involved in blood pressure decrease due to decreased respiratory rate are not yet known. Therefore the goals of this study will evaluate the chronic effect of breathing exercise guided on office and 24 hours blood pressure and analyse the chronic effect of breathing exercise guided over the autonomic function in hypertensive patients in stages 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive patients with or without use of antihypertensive drug therapy with office systolic blood pressure between 140 and 179 mmHg and / or office diastolic between 90 and 109mmHg).
* Adults over 18 years.
* Both genders.

Exclusion Criteria:

* Use of medications that alter sympathetic nerve activity (beta blockers and / or sympatholytics).
* Use of three or more classes of antihypertensive drugs
* Secondary Hypertension
* Chronic Respiratory Disease
* Diabetes Mellitus.
* Chronic Kidney Disease with Clearance Creatinine <60 ml/min
* Congestive heart failure
* Coronary disease
* Pregnant
* BMI > 30 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
blood pressure reduction | 8 weeks after the randomization
  The blood pressure reduction in mmHg will be verified by office blood pressure measurement and ambulatory blood pressure monitoring (ABPM)

SECONDARY OUTCOMES:
autonomic regulation | 8 weeks after randomization
  The autonomic function will be verified in the beginning and after 8 weeks from randomization as follows: muscle sympathetic nervous activity (MSNA) by microneurography technique (burst/min), plasma catecholamines levels (pg/ml) and heart rate variability by power spectral analysis (ms).

CONTACTS AND LOCATIONS:
Overall Officials: Decio Mion Junior, MD, Study Chair — General Hospital of School of Medicine - University of Sao Paulo
Locations (1):
- General Hospital of School of Medicine - Universiy of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Barros S, da Silva GV, de Gusmao JL, de Araujo TG, de Souza DR, Cardoso CG Jr, Oneda B, Mion D Jr. Effects of long term device-guided slow breathing on sympathetic nervous activity in hypertensive patients: a randomized open-label clinical trial. Blood Press. 2017 Dec;26(6):359-365. doi: 10.1080/08037051.2017.1357109. Epub 2017 Jul 20. PMID 28724309